CLINICAL TRIAL: NCT04399486
Title: Hemodynamic Effects of Aquatic vs. Land Exercise in Patients With Orthostatic Hypotension: a Randomized Controlled Crossover Trial
Brief Title: Hemodynamic Effects of Aquatic vs. Land Exercise in Patients With Orthostatic Hypotension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 and prolonged pool closure
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Emily Dunlap, Doctoral Student, Physical Therapist, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11-0112
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Orthostatic Hypotension
Keywords: aquatic therapy, aquatic exercise, orthostatic hypotension, blood pressure, heart rate, hemodynamics, land-based, inpatient rehabilitation,
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Physical Therapy (Experimental)
  Interventions: Other: Physical Therapy
- Land-based Physical Therapy (Active Comparator)
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical Therapy is a therapeutic exercise, education and functional activities provided on a one to one basis with a licensed Physical Therapist to meet functional goals.

SUMMARY:
Orthostatic hypotension is a highly prevalent deficit in the aging population especially when coupled with stroke, frailty, diabetes, Parkinson's disease or spinal cord injuries. This population has difficulty with the autonomic regulation of blood pressure and experiences elevated risks of falls. The fall risk is greatest when the person transitions from supine or sitting to standing as this is when blood has a tendency to pool in the legs preventing adequate blood circulation to vital organs. This is a safety concern and limiting factor for rehabilitation of patients with orthostatic hypotension in the inpatient rehabilitation setting. There is low-quality evidence that compression garments such as abdominal binders and compression stockings can be helpful to manage orthostatic hypotension and the associated fall risk. However, many people with orthostatic hypotension perceive the treatment approach with compression stockings to be largely unacceptable.

Aquatic immersion may provide better advantages to compression garments because hydrostatic pressure exerts a little over 22 mmHg pressure for every foot of water. Therefore, an individual standing in 4 ft depth water will have roughly 90 mmHg pressure on their feet and about 56 mmHg at their knees. These amounts of pressure are more than those induced by typical compression stockings, which provide 30-40 mm Hg pressure. In addition, immersion at level of xiphoid process or higher is known to translocate blood from the lower to the center of the body and act to increase cerebral blood flow which may be beneficial for preventing orthostatic hypotension symptoms.

No studies have looked at the physiologic response to immersion and aquatic exercise for people with orthostatic hypotension. Since this population is known to have difficulty with autonomic regulation of blood pressure, it is unclear if they will experience a similar hemodynamic response during immersion than the healthy population during or after aquatic therapy due to orthostatic hypotension.

Anecdotal evidence suggests that patients with orthostatic hypotension do not exhibit adverse effects due to orthostatic hypotension when standing in water or participating in aquatic exercise independent of compression garments use. They often have improved standing tolerance in the pool compared with prolonged standing on land. Steps to manage orthostatic hypotension when out of the pool, such as hydration during pool session, placing compressive garments prior to exit of pool and slow transitions out of pool setting has been adequate to prevent symptoms of orthostatic hypotension in the post exercise period in this population.

The primary aim of this study is to look at heart rate and blood pressure response when going from sit to stand during physical therapy sessions on land compared to in the pool for people who have orthostatic hypotension (defined as a drop in systolic blood pressure of at least 15 mmHg or 7 mmHg drop in diastolic blood pressure from sitting to standing). The secondary aim of this study is to evaluate tolerance for physical activity during physical therapy sessions in the pool compared to on land for people with orthostatic hypotension. The third aim of the study is to investigate heart rate and blood pressure response for 3 hours following the physical therapy sessions.

We hypothesize that orthostatic hypotension will be reduced and standing exercise tolerance will be increased when in the pool compared to on land. In addition, we hypothesized that there will not be a significant difference in heart rate or blood pressure response in the 3-hour post exercise period of aquatic vs. land exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Patient at Central Texas Rehabilitation Hospital in Austin, Texas
2. Age 18 years or older
3. Patient presents with orthostatic hypotension defined as transitions from sit to stand using a threshold of drop of at least 15 mmHg for SBP or at least 7 mmHg for DBP.
4. Aquatic therapeutic exercise is included in patients plan of care.
5. Signed informed consent

Exclusion Criteria:

1. Contraindication for aquatic physical therapy including but not limited to open wound that cannot be safely covered with a waterproof dressing, diarrhea, fever or know contagious infection.
2. Unable to safely maintain standing position for 2 min with or without assistance to measure vitals in pool and land.
3. Change in blood pressure medication or medical status between pool and land data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic variables - heart rate | up to 3 hours
  heart rate
Hemodynamic variables - blood pressure | up to 3 hours
  systolic blood pressure (SBP) and diastolic blood pressure (DBP) taken with a validated, automatic blood pressure recorder

SECONDARY OUTCOMES:
Orthostatic Hypotension symptoms | pre-post physical therapy intervention, 1 hour and 3 hours post physical therapy intervention
  Orthostatic Hypotension Questionnaire

OTHER OUTCOMES:
Characteristics of physical therapy session | during 60 min physical therapy session
  Evaluate percentage of time with sitting, standing, supine exercises vs resting.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dunlap, PT, Principal Investigator — University of Texas at Austin
Locations (1):
- Central Texas Rehabilitation Hospital, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No